CLINICAL TRIAL: NCT02086695
Title: Early Detection of Broken Hearts in Cancer Patients: Bevacizumab, Sunitinib and Heart Failure
Brief Title: Early Detection of Broken Hearts in Cancer Patients
Acronym: ASPER
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: The Asper Foundation (Unknown); St. Boniface Hospital (Other); Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Sharon Mulvagh, Consultant of Cardiology Noninvasive, Mayo Clinic
Other Study IDs: 12-005362
Record Dates: First submitted 2013-10-16; First posted 2014-03-13 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Cardiotoxicity
Keywords: Chemotherapy; Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be drawn to measure blood biomarkers to determine your heart biomarker [High sensitivity TnT and NT-proBNP] as an indicator of early heart failure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Group: All subjects with cancer who will be treated with anyone of the following chemotherapy drugs; Pazopanib, Sutent or Bevacizumab

SUMMARY:
The early detection of BVZ or Sunitinib mediated cardiotoxicity using cardiac biomarkers and novel Transthoracic Echocardiogram (TTE) techniques may allow one to adjust treatment and/or administer prophylactic cardioprotective agents, prior to the development of irreversible cardiac dysfunction. We hypothesize that cardiac biomarkers, TVI/strain-derived indices will be able to accurately detect subtle cardiac injury at a time when conventional Left Ventricular Ejection Fraction (LVEF) remains normal in BVZ or Sunitinib mediated cardiotoxicity. Additionally, we hypothesize that Endothelial Function Test (EndoPAT) testing can detect early BVZ or Sunitinib mediated endothelial dysfunction.

DETAILED DESCRIPTION:
A total of 100 individuals (50 receiving BVZ and 50 receiving Sunitinib) will be prospectively enrolled . (80 at Mayo Clinic [80 receiving BVZ, Sunitinib ,or Pazopanib] and 20 at St. Boniface General Hospital (SBGH)). Patients receiving either BVZ 5mg/kg iv ,Sunitinib 50 mg po daily, or Pazopanib for advanced Metastatic carcinoma will be screened for potential eligibility in the study. For metastatic renal cancer treatments, Sunitinib doses are (oral) 50 mg once a day for 4 weeks followed by a two week off period. The six week cycle is then repeated. In case of toxicities observed with the dose, a 25% reduction in the daily dose during the "on" period is performed (37.5 mg). Patients will be studied at 7 time points: i) Baseline; ii) Day 1; iii) Day 5; iv) 4-6 weeks ; v) 3 months; vi) 6 months after the initiation of both drugs (BVZ and Sunitinib) ; and vii) 12 months after the initiation of BVZ drug only (Figure 1). Three visits (baseline, 4-6 weeks , and 3 months) are considered part of standard clinical care, and four visits are for research. At each visit, in addition to standard of care provided by the Oncologist, blood will be drawn to measure high sensitivity troponin-T (hsTnT) and Natriuretic-proBNP. The patients will also undergo a TTE with tissue velocity imaging (TVI), strain and left ventricular opacification (LVO) and myocardial perfusion at each time point. EndoPAT test will also be performed at baseline, and 3 months. The baseline, 4-6 weeks, and 3 month visits will be part of your standard clinical care and followup.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer
2. Treatment plan includes BVZ ,Sunitinib, or Pazopanib
3. Ages 18 - 90 years old -

Exclusion Criteria: Left Ventricular EF < 50%

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 individuals with advanced metastatic renal cell carcinoma or colorectal cancer (50 receiving BVZ and 50 receiving Sunitinib) will be prospectively enrolled . (80 at Mayo Clinic( Any subject presenting who will be treated for cancer recieving Pazopanib, Sutent, or Bevacizumab] and 20 at St. Boniface General Hospital (SBGH)).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with changes in Tissue velocity imaging (TVI), myocardial deformation indices (Strain, strain rate, twist and torsion), and diastolic function indices (Mitral Valve Pulsed Wave Doppler, Tissue Doppler Imaging, Left Atrial volumes) | Baseline to 2 years

SECONDARY OUTCOMES:
Number of participants with changes in quantitative myocardial perfusion parameters including myocardial blood flow velocity and myocardial blood flow derived from contrast perfusion echocardiography | Baseline to 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No